CLINICAL TRIAL: NCT05697978
Title: Distance and Intermediate Visual Acuity in Patients With Implanted Monofocal Negative Aspheric Intraocular Lens
Acronym: CLAINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Očni centrum Praha a.s. (Unknown); Somich, s.r.o. (Other)
Responsible Party: Principal Investigator, Andrea Janekova, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZ-001
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Intraocular Lens
Keywords: intraocular lens; monofocal lens; intermediate visual acuity

STUDY DESIGN:
Intervention Model Description: each patient in group received monofocal intraocular lens in both eyes
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monofocal lens (Other): Eyes of patients with implanted monofocal aspheric lens Clareon (Alcon LLC)
  Interventions: Device: Monofocal intraocular lens Clareon (Alcon LLC)

INTERVENTIONS:
Device: Monofocal intraocular lens Clareon (Alcon LLC) — monofocal aspheric lens implanted in eyes of patient during routine cataract surgery

SUMMARY:
To get the visual outcomes for distance and intermediate and binocular defocus curve in patients with implanted monofocal intraocular lens Clareon (IOL; model SY60CL; Alcon Vision LLC) at 3 months after the surgery.

DETAILED DESCRIPTION:
The goal of refractive cataract surgery is to remove the opacity, or cataract and to produce the desired refractive outcome. In most cases, the desired outcome is an emmetropic eye, or an eye that sees 20/20 Snellen for distance vision post-surgery with the implant of a monofocal IOL. This, however, does not offer much in the way of intermediate and near vision. The increased desire for simultaneous distance, intermediate and near vision has increased the popularity of multifocal IOLs (MIOLs). However MIOLs provide visual acuity for all distances, they has occurence of optical phenomena such as glare and halo and lower contrast sensitivity. Extended depth of focus (EDOF) lens should provide distance vision as good as monofocal lens and intermediate vision better than monofocal but without or with less appearance of optical phenomenon or decreased contrast sensitivity.

This study is prospective, multi-center, conducted from 10/2022 to 08/2023 in the Ophthalmology department of Faculty Hospital Kralovske Vinohrady in Prague, in Eye Center Prague and Eye Clinic SOMICH (Karlovy Vary). The research protocol was explained to all participants and informed consent was signed before enrolling patient to the study. The study was approved by the Ethics Committee of Faculty Hospital Kralovske Vinohrady and will enrolled up to 100 patients with presence of cataract in both eyes.

Bilateral clear corneal phacoemulsification and IOL implantation is performed by two experienced surgeon using the same technique in both eyes. The surgical process involved topical anesthesia, superior 3-step clear corneal incision (2,2mm), 5,0mm curvilinear capsulorhexis, phacoemulsification, bilateral irrigation- aspiration and implantation of monofocal aspheric intraocular lens (Clareon Alcon vision LLC).

Patients are scheduled for visit at 3 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* presence of cataract in both eyes
* no other ocular pathology affecting visual acuity
* bilateral phacoemulsification cataract surgery was arranged for both eyes
* corneal astigmatism up to 0,5 cylinder (measured by IOL Master biometry)
* dioptric power of both selective lens within 1,5 D range in one patient
* selecting IOL power between 15 D and 28 D power range

Exclusion Criteria:

* complicated cataract
* corneal opacities or irregularities
* amblyopia
* anisometropia
* coexisting ocular pathologies
* glaucoma
* history of ocular surgery
* refusal or unable to maintain follow-up

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Monocular corrected Distance Visual Acuity (CDVA) | 3 months
  Monocular corrected distance visual acuity (CDVA) is measured at 4 m using an ETDRS (Early Treatment Diabetic Retinopathy Study) illumination cabinet (Precision Vision) under photopic conditions.
Binocular corrected Distance Visual Acuity (CDVA) | 3 months
  Binocular corrected distance visual acuity (CDVA) is measured at 4 m using an ETDRS (Early Treatment Diabetic Retinopathy Study) illumination cabinet (Precision Vision) under photopic conditions.
Monocular uncorrected intermediate visual acuity (UIVA) | 3 months
  Monocular intermediate visual acuity is measured using printed ETDRS charts for distance of 66cm
Binocular uncorrected intermediate visual acuity (UIVA) | 3 months
  Binocular intermediate visual acuity is measured using printed ETDRS charts for distance of 66cm
Monocular distance corrected intermediate visual acuity (DCIVA) | 3 months
  Monocular distance corrected intermediate visual acuity is measured using printed ETDRS charts for distance of 66cm
Binocular distance corrected intermediate visual acuity (DCIVA) | 3 months
  Binocular distance corrected intermediate visual acuity is measured using printed ETDRS charts for distance of 66cm

SECONDARY OUTCOMES:
Binocular defocus curve | 3 months
  A defocus curve that measures visual acuity should be obtained by using the best corrected distance refraction and then defocusing the image in 0.5 increments from +1.5 to -3.0 diopter with spherical plus and spherical minus trial lenses (i.e.,+1.5 D, +1.0 D, +0.5 D, 0.00 D, -0.5 D, -1.00 D, . . . ,-2.50 D) with visual acuity recorded at each change in correction.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Janekova, MD, Principal Investigator — Eye Center Prague
Locations (3):
- Czechia (3):
  - Eye Center Prague, Prague, Czech Republic
  - Faculty hospital Kralovske Vinohrady, Prague, Czech Republic
  - Somich Eye Clinic, Karlovy Vary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lehmann R, Maxwell A, Lubeck DM, Fong R, Walters TR, Fakadej A. Effectiveness and Safety of the Clareon Monofocal Intraocular Lens: Outcomes from a 12-Month Single-Arm Clinical Study in a Large Sample. Clin Ophthalmol. 2021 Apr 20;15:1647-1657. doi: 10.2147/OPTH.S295008. eCollection 2021. PMID 33907378
- [Result] Werner L, Thatthamla I, Ong M, Schatz H, Garcia-Gonzalez M, Gros-Otero J, Canones-Zafra R, Teus MA. Evaluation of clarity characteristics in a new hydrophobic acrylic IOL in comparison to commercially available IOLs. J Cataract Refract Surg. 2019 Oct;45(10):1490-1497. doi: 10.1016/j.jcrs.2019.05.017. Epub 2019 Aug 6. PMID 31399323
- [Result] Bala C, Poyales F, Guarro M, Mesa RR, Mearza A, Varma DK, Jasti S, Lemp-Hull J. Multicountry clinical outcomes of a new nondiffractive presbyopia-correcting IOL. J Cataract Refract Surg. 2022 Feb 1;48(2):136-143. doi: 10.1097/j.jcrs.0000000000000712. PMID 34288635